CLINICAL TRIAL: NCT00707902
Title: Multicentric Randomized Double Blind Double Dummy Placebo Controlled Clinical Trial for Assessment of Safety and Efficacy of a Echinacea/Sage Spray in Comparison to a Chlorhexidine/Lidocaine Spray in the Treatment of Acute Sore Throats
Brief Title: Clinical Trial for Assessment of Safety and Efficacy of a Echinacea/Sage Spray Compared to a Chlorhexidine/Lidocaine Spray in the Treatment of Acute Sore Throats
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Responsible Party: Andy Suter, Head of Medical Dept., Bioforce AG, Roggwil, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 920'073
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2008-07-01 (Estimated); Status verified 2008-06

CONDITIONS: Pharyngitis
Keywords: Sore throats,; Pharyngitis; Acute
MeSH Terms: conditions — Pharyngitis | interventions — chlorhexidine gluconate, lidocaine drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Drug: Echinacea/sage
  patients received additionally a placebo-spray for the synthetical comparator (chlorhexidine/lidocaine) as the study was double dummy blinded.
  Patients had to apply spray every 2 hours with two puffs to the pharyngeal area up to a maximum of 10 times daily. Treatment duration was until illness was resolved or for a maximum of 5 consecutive days.
  Arms: 1
  Interventions: Drug: echinacea/sage
- 1 (Active Comparator): Drug: Chlorhexidine/lidocaine
  patients received additionally a placebo-spray for the synthetical comparator (echinacea/sage) as the study was double dummy blinded.
  Patients had to apply spray every 2 hours with two puffs to the pharyngeal area up to a maximum of 10 times daily. Treatment duration was until illness was resolved or for a maximum of 5 consecutive days.
  Interventions: Drug: chlorhexidine/lidocaine

INTERVENTIONS:
Drug: chlorhexidine/lidocaine
  Arms: 1
Drug: echinacea/sage
  Arms: 2

SUMMARY:
The aim of the study is to show non-inferiority of an echinacea/sage spray compared to a chlorhexidine/lidocaine-spray in the treatment of acute sore throat during five days of treatment.

Main outcome parameter is the non-inferiority in number of responders between the two treatment groups. A responder is defined as a reduction by 50% of the total baseline score taken prior to treatment start. The symptoms are assessed with a symptom score.

DETAILED DESCRIPTION:
Further secondary parameters are :

Responders during at day 4 and 5, single symptom scores during 1 to 5 days of observation, pain at begin and end (100mm VAS), assessment of efficacy by physician and patient, consumption of rescue medication

Assessment of safety by physician and patient, frequency of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Age > 12 years;
* Acute pharyngitis or tonsillitis with symptoms of throat pain and inflammation of the pharynx and/or tonsils;
* Onset of sore throat less than 72 hours before inclusion ;
* A Tonsillopharyngitis Severity Score ≥6;
* Written informed consent.

Exclusion Criteria:

* Analgesics <12 hours;
* Antibiotics <24 hours; t
* Topical throat pain medication <4 hours;
* Systemic corticosteroids within the last month;
* Symptoms of primary bacterial pharyngitis or secondary bacterial infection;
* Serious illness such as tumors; allergy to one of the ingredients; pregnancy or lactation;
* Hypersensitivity to ibuprofen;
* Participation in another clinical trial in the previous 30 days.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2006-02; Study Completion 2006-08

PRIMARY OUTCOMES:
comparison of responder of the two treatment groups after the first, second, and third days. A responder is defined as a reduction by 50% of the total baseline score taken prior to treatment start. | first three days of treatment

SECONDARY OUTCOMES:
Comparison of response rates after 4th and 5th days of treatment; VAS throat pain; amount rescue medication used; global assessment efficacy Frequency of adverse events, global assessment of tolerability | five days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Kähler, MD, Principal Investigator — General practice, Hubstrasse 37, 9500 Wil, Switzerland
Locations (1):
- Allergy Clinic, Landquart, Switzerland

REFERENCES:
- [Result] Gertsch J, Schoop R, Kuenzle U, Suter A. Echinacea alkylamides modulate TNF-alpha gene expression via cannabinoid receptor CB2 and multiple signal transduction pathways. FEBS Lett. 2004 Nov 19;577(3):563-9. doi: 10.1016/j.febslet.2004.10.064. PMID 15556647
- [Result] Shah SA, Sander S, White CM, Rinaldi M, Coleman CI. Evaluation of echinacea for the prevention and treatment of the common cold: a meta-analysis. Lancet Infect Dis. 2007 Jul;7(7):473-80. doi: 10.1016/S1473-3099(07)70160-3. PMID 17597571
- [Result] Bereznoy VV, Riley DS, Wassmer G, Heger M. Efficacy of extract of Pelargonium sidoides in children with acute non-group A beta-hemolytic streptococcus tonsillopharyngitis: a randomized, double-blind, placebo-controlled trial. Altern Ther Health Med. 2003 Sep-Oct;9(5):68-79. PMID 14526713
- [Result] Hubbert M, Sievers H, Lehnfeld R, Kehrl W. Efficacy and tolerability of a spray with Salvia officinalis in the treatment of acute pharyngitis - a randomised, double-blind, placebo-controlled study with adaptive design and interim analysis. Eur J Med Res. 2006 Jan 31;11(1):20-6. PMID 16504956
- [Derived] Schapowal A, Berger D, Klein P, Suter A. Echinacea/sage or chlorhexidine/lidocaine for treating acute sore throats: a randomized double-blind trial. Eur J Med Res. 2009 Sep 1;14(9):406-12. doi: 10.1186/2047-783x-14-9-406. PMID 19748859